CLINICAL TRIAL: NCT01007357
Title: Abdominal MR Imaging at 3.0T: Sequence Optimization and Implementation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left institution; did not complete the study
Sponsor: University of Nebraska (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0290-09-FB
Record Dates: First submitted 2009-10-28; First posted 2009-11-04 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Diffuse and Focal Abnormalities of the Liver and Pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body MRI healthy volunteers (Other): Body MRI to optimize sequences in healthy individuals and in disorder subjects
  Interventions: Device: Body MR imaging

INTERVENTIONS:
Device: Body MR imaging — Body MR imaging will be performed to optimize sequences
  Other Names: Body MR imaging performed to optimize sequences

SUMMARY:
This project will facilitate the optimization of body MR imaging at 3 Tesla.

DETAILED DESCRIPTION:
This project is meant to improve the image quality of multiple sequences at 3.0T applied to the abdominal and pelvic regions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ages of 19 and 65
* Healthy volunteer subjects should not have any history of disease or symptoms - based on clinical history
* Subjects with an underlying disorder (diffuse and focal abnormalities of the liver and pancreas)

Exclusion Criteria:

* Inability to provide informed consent
* A medical or contraindications that will prevent subjects from having a MRI
* Subjects with severe renal dysfunction or patients on dialysis

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12-15 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Optimizing body MR imaging sequences | 2 years
  Healthy volunteers will be used to obtain optimized body MR imaging sequences that will then be used to evaluate MR imaging sequences of subjects with underlying disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Hussain, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States